CLINICAL TRIAL: NCT06521762
Title: Etrasimod for Immune Checkpoint Inhibitor Diarrhea and Colitis
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early as no patients were enrolled.
Sponsor: Yale University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Harriet Kluger, Harvey and Kate Cushing Professor of Medicine (Oncology) and of Dermatology, Yale University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2000036896
Record Dates: First submitted 2024-07-21; First posted 2024-07-26 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Immune Checkpoint Inhibitor-Related Diarrhea and Colitis
MeSH Terms: conditions — Colitis | interventions — etrasimod; Adrenal Cortex Hormones

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Etrasimod plus corticosteroids (Experimental): Participants will receive Etrasimod plus corticosteroids, to be given up to 120 days, to treat IMDC.
  Interventions: Drug: Etrasimod; Drug: Corticosteroids
- Placebo plus corticosteroids (Placebo Comparator): Participants will receive Placebo plus corticosteroids, to be given up to 120 days, to treat IMDC.
  Interventions: Drug: Placebo; Drug: Corticosteroids

INTERVENTIONS:
Drug: Etrasimod — 2 mg/day oral tablet
  Other Names: VELSIPITY
  Arms: Etrasimod plus corticosteroids
Drug: Placebo — matching placebo oral tablet
  Arms: Placebo plus corticosteroids
Drug: Corticosteroids — Corticosteroids will be given in conjunction with study drug or placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, two-arm phase 2 study of etrasimod plus corticosteroids versus placebo plus corticosteroids for the treatment of IMDC CTCAE v5.0 grade ≥ 2 due to ICI therapy alone (α-PD-(L)1 monotherapy or combined with another ICI, such as α-CTLA-4 or α-LAG-3) or ICI plus an oral tyrosine kinase inhibitor that in the opinion of the treating physician requires treatment with corticosteroid-based immunosuppression and does not require immediate secondary immune suppression, such as vedolizumab or infliximab (or equivalent).

IMDC is one of the most common Immune Related Adverse Events (irAEs) from treatment with ICI. Current guidelines recommend steroid treatment for IMDC CTCAE grade ≥ 2, which requires temporary or permanent cessation of ICI therapy. Corticosteroids may interfere with the anti-tumor activity of ICIs and are therefore not co-administered. Strategies are needed to both reduce the dose and duration of corticosteroids needed for IMDC treatment and minimize the duration off ICI therapy before re-administering ICI (for those patients in whom it is deemed safe to rechallenge).

DETAILED DESCRIPTION:
Participants will be screened as soon as IMDC is suspected but will not be randomized and administered the first dose of etrasimod or placebo until results from Clostridium difficile (C. difficile) and other intestinal infection assays are confirmed to be negative and stool calprotectin confirmed to be positive. If intestinal infectious studies are positive the participant will be excluded from the study. Due to the acute nature of some cases of IMDC (e.g., grade 4 IMDC), some participants may require initiation of corticosteroids before enrollment. In these cases, participants may be enrolled if the first dose of etrasimod or placebo can be administered within 96 hours of the first dose of corticosteroids. Participants will undergo flexible sigmoidoscopy or colonoscopy with colon biopsy prior to, within the first 7 days of starting study drug, which will be repeated 7 to 14 days after completing the last dose of study drug.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced unresectable or metastatic cancer
* Any tumor type being treated with either α-PD-(L)1 monotherapy or combination therapy containing α-PD-(L)1 and another ICI such as α-CTLA-4 or α-LAG-3 therapy.
* Patients receiving ICI(s) in combination with oral tyrosine kinase inhibitors (TKIs) may be enrolled if their diarrhea persists despite holding the TKI for 5 days and they meet the other eligibility criteria. These cases should be discussed with one of the study PIs. Patients receiving chemotherapy in combination with ICI(s) cannot be enrolled.
* Grade ≥ 2 IMDC requiring immunosuppression with corticosteroids as defined by at least grade 2 diarrhea and grade 2 colitis by CTCAE v5.0, which are defined in Appendix 3 (section 11.3) of the protocol.
* Positive stool calprotectin test
* Able to provide informed consent.
* Able and willing to take the study medication and comply with all study requirements.
* The following medical criteria are met:

  1. No known history of inflammatory bowel disease
  2. Vital signs at screening: pulse rate ≥ 50 beats per minute, systolic blood pressure ≥ 90 mm Hg, and diastolic blood pressure ≥ 55 mm Hg
  3. 12-lead electrocardiogram (ECG) that showed no clinically significant abnormalities as defined by the clinician's judgement at the time the ECG was performed
* Healthcare professional-confirmed history of varicella or a full course of vaccination against varicella zoster virus (VZV) or a positive antibody test to VZV
* Eligible patients that were biologically female at birth must be:

  1. Non-pregnant, as determined by qualitative urine hCG testing
  2. Non-lactating
  3. If premenopausal, be either surgically infertile OR using 2 acceptable methods of birth control for 30 days after the last dose of etrasimod is administered (inquire for a list of birth control methods considered acceptable)

Exclusion Criteria

* Patients receiving ICIs in the adjuvant setting.
* Patients with severe hepatic impairment, as indicated by having a Child-Pugh C score.
* The following infectious complications:

  1. difficile infection, or an intestinal bacterial or parasitic infection detected by a multiplexed stool infection assay
  2. Have received treatment for C. difficile infection within 30 days or another intestinal pathogen within 30 days prior to enrollment
  3. Have a known history of active or latent tuberculosis, or active hepatitis B or hepatitis C
  4. Have a known history of congenital or acquired immunodeficiency, including but not limited to common variable immune deficiency (CVID) and human immunodeficiency virus (HIV) infection
  5. Have evidence of abdominal abscess or toxic megacolon at the initial screening visit
* Patients with diabetes mellitus that meet the following criteria:

  1. Type 1 diabetes mellitus
  2. Uncontrolled type 2 diabetes mellitus requiring insulin for routine management
* Have a history of severe respiratory disease (i.e., pulmonary fibrosis, asthma, and chronic obstructive pulmonary disease) requiring supplemental oxygen not related to an underlying malignancy
* Have the following cardiovascular history:

  1. In the last 6 months, experienced myocardial infarction, unstable angina pectoris, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or Class III or IV heart failure.
  2. Unstable ischemic heart disease, Class I or II heart failure, history of cardiac arrest, cerebrovascular disease, or uncontrolled hypertension, unless consulting cardiologist believes safe
  3. History or presence of Mobitz type I or II second-degree, or third-degree atrioventricular (AV) block, sick sinus syndrome, or sino-atrial block, unless the patient has a functioning pacemaker.
  4. A history or presence of recurrent symptomatic bradycardia or recurrent cardiogenic syncope, or severe untreated sleep apnea
  5. QTcF interval ≥ 450 ms in men or ≥ 470 ms in women
  6. Arrhythmias requiring treatment with Class Ia or Class III anti-arrhythmic drugs or QT prolonging drugs, unless consulting cardiologist believes safe
* Have received treatment that could be considered secondary IMDC treatment within 4 half-lives of the agent, including but not limited to vedolizumab, anti-TNFα antibodies, and mycophenolate mofetil. Treatments that could be considered secondary IMDC treatment but are not specified in this protocol will be adjudicated by a study PI or co-PI at the time of screening.
* Have a known history of macular edema
* Have a history of any clinically significant medical condition that, in the investigator's opinion, precludes participation in the study
* History of an opportunistic infection (e.g., Pneumocystis jirovecii, cryptococcal meningitis, progressive multifocal leukoencephalopathy) or history of disseminated herpes simplex or disseminated herpes zoster.
* Have an absolute neutrophil count (ANC) or absolute lymphocyte count (ALC) < 500
* Have received any investigational therapy, excluded medications (Appendix 4, section 11.4), or any approved therapy in an investigational protocol within 14 days before screening.
* Have active psychiatric problems that, in the investigator's opinion, could interfere with compliance with the study procedures.
* Have been using moderate to strong inhibitors of cytochrome P450 (CYP)2C9.
* Unable to discontinue any of the drugs listed in Appendix 4 (section 11.4) of the protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Average daily weight-adjusted dose of corticosteroids use | up to day 120 or when a censoring event occurs
  Average daily weight-adjusted dose of corticosteroids use (up to day 120 or when a censoring event occurs), accounting for both the weight-adjusted cumulative dose of steroids and the length of treatment.

SECONDARY OUTCOMES:
Requirement for secondary immunosuppression | up to day 120 or when a censoring event occurs
  Requirement for secondary immunosuppression throughout the study period (up to day 120 or when a censoring event occurs), a binary variable (Yes or No). Numbers of participants that answered Yes/No.
Mean time to improvement | up to day 120 or when a censoring event occurs
  Mean time to first improvement to CTCAE v5.0 grade ≤ 1 for IMDC in days
Mean number of days without corticosteroids use | up to day 120 or when a censoring event occurs
  Mean number of days without corticosteroids use
Safety and Tolerability Measured by Assessing Incidence and severity of adverse events of special interest. | up to day 120 or when a censoring event occurs
  Incidence and severity of adverse events of special interest. Number of participants that experience any adverse event of special interest determined by CTCAE v5.0.
Incidence and severity of laboratory abnormalities | up to day 120 or when a censoring event occurs
  Incidence and severity of laboratory abnormalities. Total count of clinically significant abnormal labs, determined by CTCAE
Total count of clinically significant vital sign abnormalities | up to day 120 or when a censoring event occurs
  Count of clinically significant vital sign abnormalities

CONTACTS AND LOCATIONS:
Overall Officials: Harriet Kluger, MD, Principal Investigator — Yale University
Locations (1):
- Yale Cancer Center, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No